CLINICAL TRIAL: NCT05960058
Title: Acceptance and Effectiveness of SARS-COV-2 Vaccination in Systemic Sclerosis Patients Treated by Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Acceptance and Effectiveness of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2) Vaccination in Systemic Sclerosis Patients Treated by Autologous Hematopoietic Stem Cell Transplantation
Acronym: COV2-VACCinSSc
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230473
Record Dates: First submitted 2023-07-24; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Systemic Sclerosis; SARS-CoV 2 Vaccination
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases (Autologous Haematopoietic Stem Cell Transplantation (AHSCT)): Systemic Sclerosis (SSc) patients treated by AHSCT and actively followed at Saint Louis on January 1st, 2021
- Controls (without Autologous Haematopoietic Stem Cell Transplantation): Systemic Sclerosis (SSc) patients treated by AHSCT and actively followed at Saint Louis on January 1st, 2021

SUMMARY:
On December 27th 2020, the implementation of SARS-CoV-2 vaccination in France first became available amongst all immunosuppressed patients at very high risk of severe Coronavirus Disease (COVID-19) infection, specifically for Hematopoietic Stem Cell Transplant recipients or other fragile immunosuppressed patients.

Systemic sclerosis (SSc) is an autoimmune disease characterized by dysregulation of the immune system, vascular damage and progressive fibrosis of the skin and internal organs (heart, lung and kidney) which may lead to severe comorbidities and SSc-related mortality. In severe rapidly progressive SSc, we and others demonstrated that autologous hematopoietic stem cell transplantation (AHSCT) is the only treatment so far allowing improvement in overall and event free survival up to 7 years after AHSCT.

As soon as vaccines were available on January 1st, 2021 and following the French Haute Autorité de Santé (HAS) and Société Francophone de Greffe de Moelle et de Thérapie Cellulaire (SFGM-TC) good clinical practices (GCP) guidelines, the ad hoc COVID19 vaccinations were proposed to all SSc patients in France, including those previously treated by AHSCT and followed at Maladies Auto Immunes et Thérapie Cellulaire (MATHEC) Center of Reference for stem cell therapy at St-Louis hospital. In July 2021, the Autoimmune Diseases Working Party (ADWP) and the European society for Blood and Marrow Transplantation (EBMT) guidelines recommended vaccination against SARS-CoV2 as early as 3 months after HSCT for autoimmune diseases.

Only one Israeli study so far has analyzed the efficacy of SARS-CoV-2 vaccination after autologous HSCT (AHSCT) in SSc patients..

We therefore designed the present case control study retrospective study to assess the acceptance and effectiveness of this vaccination program in SSc patients treated by AHSCT as compared to other fragile SSc individuals.

The Primary objective is to evaluate the effectiveness of implementing the anti-SARS-CoV2 vaccination program according to the French GCP for COVID-19 prophylaxis in SSc fragile patients, in terms of risk of asymptomatic or symptomatic COVID-19 infection, among SSc patients treated by AHSCT compared to 1:1 matched non transplant SSc controls.

ELIGIBILITY:
Inclusion Criteria:

1. Adults SSc patients fulfilling criteria from the American College of Rheumatology- European League Against Rheumatism for systemic sclerosis, the 1980 criteria from the American College of Rheumatology for systemic sclerosis
2. SSc patients who were offered SARS-CoV-2 vaccination program according to French GCP (with at least either a two-dose mRNA vaccine or single-dose adenoviral vector) between Jan 1st 2021 to June 30th 2022
3. a) Cases: SSc patients, actively followed on Jan 1st 2021 and who underwent treatment by AHSCT therapy from 1998 up to December 31st 2020 b) Controls (non AHSCT): SSc patients, actively followed on Jan 1st 2021 and who had not undergone treatment by AHSCT at that time nor up to June 30th 2022
4. Informed patients followed at Filière des maladies Auto-immunes et Auto Inflammatoires Rares (FAI2R) systemic sclerosis centers: either Centre de Référence des Maladies Rares (CRMR) MATHEC, Maladies Auto-immunes et Thérapie Cellulaire" at Saint-Louis hospital (Paris) or from "Service de Médecine Interne et Immunologie Clinique" at Rangueil hospital (Toulouse).

Exclusion Criteria:

1. SSc patient who were opposed to their data analysis after information about the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Systemic Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of asymptomatic or symptomatic COVID-19 infection after AHSCT as compared to non AHSCT SSc patients. | Up to 18 months
  Asymptomatic COVID-19 are defined by positive Polymerase Chain Polymerase (PCR) on routine testing (contact case or fortuitous discovery). Symptomatic COVID-19 patients are defined by positive PCR test and clinical symptoms related to COVID-19 infection.

SECONDARY OUTCOMES:
Proportion of SSc patients, previously treated by AHSCT and in non-transplant controls, who refused vaccination during the study period | Up to 18 months
Cumulative incidence of symptomatic COVID-19 infection in SSc patients previously treated by AHSCT and in non-transplant controls | Up to 18 months
Time of onset of first COVID-19 infection (symptomatic or asymptomatic) diagnosed during the study period after completing at least 2 vaccines injections in SSc patients previously treated by AHSCT and in non-transplant controls | Up to 18 months
Severity of symptomatic COVID-19 | Up to 18 months
  It is assessed and classified according to the care needed for each patient: asymptomatic; mild=ambulatory; moderate=hospitalised out of Intensive Care Unit (ICU); and severe=ICU or deceased
Proportion of SSc patients with at least 1 grade≥3 adverse event after COVID19 vaccination | Up to 18 months
  It is assessed according to Common Terminology Criteria for Adverse Events (CTC-AE v5.0)
Humoral response in SSc patients treated by AHSCT and in controls after messenger RiboNucleic Acid (mRNA) vaccine against SARS-CoV | Up to 18 months
  It is assessed as positive or negative, according to the presence of SARS-CoV-2 S1/S2 Immunoglobulin G (IgG) antibodies on serological test performed after the second vaccine dose or after 1 vaccine and one COVID-19 infection. Patients were considered positive or negative for being able to mount a humoral response according to national GCP guidelines (last update March 2022).The threshold for a positive immunogenic response was defined by local laboratory standards according to the manufacturer's instructions for cut-off values.

IPD SHARING:
Plan to Share IPD: Undecided